CLINICAL TRIAL: NCT06348680
Title: The Effect of Video-assisted Episiotomy Repair Training on Anxiety and Self-efficacy Levels in Midwifery Students: a Randomized Controlled Study
Brief Title: The Effect of Video-assisted Episiotomy Repair Training on Anxiety and Self-efficacy Levels in Midwifery Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AmasyaU-betuluzun-004
Record Dates: First submitted 2024-03-25; First posted 2024-04-05 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Episiotomy Wound
Keywords: Episiotomy; Self-efficacy; Midwifery Students

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Standard episiotomy repair training will be given to the students in the experimental group using the calf tongue simulator. After the theoretical phase is completed, the implementation phase will begin. During the application period (practical phase), students in this group will be shown a 'video recording' of episiotomy repair prepared by the researchers as educational material. Thus, students in the experimental group will be able to watch episiotomy repairs whenever and however many times they want, in addition to researcher support throughout the application, and improve their application skills.
  Interventions: Other: Video assisted episiotomy repair training
- Control group (No Intervention): Students in the control group will be given standard episiotomy repair training using the calf tongue simulator. After the theoretical phase is completed, the implementation phase will begin. Researcher support will be provided throughout the implementation period.

INTERVENTIONS:
Other: Video assisted episiotomy repair training — Midwifery Intervention The 'video recording' prepared by researchers specialized in the field of midwifery to increase the episiotomy repair skills of midwifery students will be used as training material. The content of the video recording is as follows: control before episiotomy repair, episiotomy repair, subcutaneous suturing, skin suturing, suturing techniques (Continuous, Simple Intermittent, Mattress). After the video recording is completed, it will be restarted and shown to the students in the experimental group continuously throughout the application period. At the end of the application period, students will be re-evaluated.
  Arms: Experimental group

SUMMARY:
The goal of midwifery undergraduate education is; To provide students with basic professional knowledge, skills and attitudes in cognitive, affective and psychomotor dimensions. Various practices are used to provide students with midwifery skills. Case studies, maintenance processes, laboratory applications, field studies, simulation application and video monitoring are some of these applications. Each of these approaches, which are especially preferred in applied courses, has an important place in increasing students' self-efficacy and reducing their anxiety. Episiotomy is one of the obstetric interventions that negatively affects the self-efficacy of midwifery students and causes anxiety. Midwives are responsible for performing and caring for episiotomy. In many countries, episiotomy repair training is given to midwifery students using sponges or models. However, today the use of calf tongue, which is very similar to perineal tissue, has become widespread. There are a limited number of studies in the literature using calf tongue simulation. These studies suggested that the practice improved the skills of midwifery students. No study has been found in the literature using video-assisted episiotomy repair training.

DETAILED DESCRIPTION:
Episiotomy is one of the most commonly performed surgical interventions in normal vaginal birth. Episiotomy, also known as perineotomy, can be defined as an incision made in the perineum to ensure easy delivery of the fetus, shorten the active phase of labor, prevent lacerations, and protect the perineal tissue and anal sphincter. This procedure is a surgical intervention applied to the bulbo-cavernos muscle located in the perineum in the second phase of labor. It can be said that episiotomy has become widespread as a result of medicalization in birth, as in all areas of health. In particular, moving births from homes to hospital environments can be cited as one of the leading reasons for the increase in episiotomy rates. Routine episiotomy may cause pelvic organ prolapse and damage the muscles in the anal sphincters and perineal structure. In addition, studies on the subject have shown that episiotomy may be associated with problems such as postpartum pain, dyspareunia and incontinence. It is also known that the rate of perineal trauma is high in countries where episiotomy is frequently performed. For this reason, episiotomy, which is basically done to prevent uncontrolled damage that may occur in the perineal area, is not routinely preferred today. The recommendation of the American College of Obstetricians and Gynecologists (ACOG) regarding episiotomy is as follows: Episiotomy may be preferred in cases of risk arising from the mother or the baby, such as protecting against perineal tears that may occur in the mother during vaginal birth, facilitating or accelerating birth, but its use should be limited in cases where it is not necessary.

Self-efficacy is defined as the individual's beliefs about his ability to perform significantly in events that will affect his life. Self-efficacy perception determines how individuals feel, think, motivate themselves and behave. It is known that motivation increases as the level of self-efficacy increases). It has also been reported that individuals with high self-efficacy have a higher potential to cope with problems, experience less stress and anxiety, and make more effort to achieve their desired results. It is estimated that people with low self-efficacy often experience stress, anxiety and depression, and their academic and social success decreases. As a matter of fact, some studies have found that the academic performance of university students increases in parallel with their self-efficacy score averages.

The goal of midwifery undergraduate education is; To provide students with basic professional knowledge, skills and attitudes in cognitive, affective and psychomotor dimensions. Various practices are used to provide students with midwifery skills. Case studies, maintenance processes, laboratory applications, field studies, simulation application and video monitoring are some of these applications. Each of these approaches, which are especially preferred in applied courses, has an important place in increasing students' self-efficacy and reducing their anxiety. Episiotomy is one of the obstetric interventions that negatively affects the self-efficacy of midwifery students and causes anxiety. Midwives are responsible for performing and caring for episiotomy. In many countries, episiotomy repair training is given to midwifery students using sponges or models. However, today the use of calf tongue, which is very similar to perineal tissue, has become widespread. There are a limited number of studies in the literature using calf tongue simulation. These studies suggested that the practice improved the skills of midwifery students. No study has been found in the literature using video-assisted episiotomy repair training.

ELIGIBILITY:
Inclusion Criteria:

* Midwifery students who are studying in the 3rd year, have taken the normal birth and postpartum period course and are registered for the risky birth and postpartum period course
* Those who volunteer to participate in the study

Exclusion Criteria:

* Those who did not agree to participate in the research
* Those who have an active working life as midwives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
State Anxiety Scale | through study completion, an average of 1 year
  Scoring is as follows: "1=Not at all, 2=Somewhat, 3=A lot and 4=Completely." There are two types of expressions in the scale: direct and reverse. Items 1, 2, 5, 8, 10, 11, 15, 16, 19, 20 are scored in reverse. Direct expressions express negative emotions; Inverted expressions contain positive emotions. The scores obtained from the scale theoretically range between 20 and 80. High scores from the scale indicate high anxiety level, low scores indicate low anxiety level.
Episiotomy Skills Self-Efficacy Scale | through study completion, an average of 1 year
  The scale consists of 19 items and two subscales: 'episiotomy preparation and application' and 'episiotomy control'. For each item on the Likert-type scale, "1" is given for the "strongly disagree" response, "2" is given for the "disagree" response, "3" is given for the "agree" response, and "4" is given for the "strongly agree" response. There are no reverse coded items in the scale. The total score varies between 19 and 76. High scores from the scale indicate a high level of self-efficacy for episiotomy skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No